CLINICAL TRIAL: NCT01297972
Title: Bone Marrow Mesenchymal Stem Cells in the Treatment of Refractory Severe Acquired Aplastic Anemia
Brief Title: Mesenchymal Stem Cells in the Treatment of Relapsed/Refractory Severe Acquired Aplastic Anemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Diego Villa Clé, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONEP 16119
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia; Mesenchymal Stem Cells
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Intravenous bone marrow mesenchymal stem cells infusion — After standard immunosuppressive therapy with rabbit antithymocyte globulin 3,5 mg/Kg/day during 5 days, allogeneic unrelated bone marrow derived mesenchymal stem cells will be infused intravenously. Oral cyclosporine 5 mg/Kg/day (with dose correction weekly to keep serum cyclosporine level between 150-250 mg/dl) up to 6 months will be added.

SUMMARY:
Mesenchymal stem cells have been tested in many autoimmune disorders with encouraging results and may be an alternative to the treatment of immune-mediated severe acquired aplastic anemia.

DETAILED DESCRIPTION:
Acquired aplastic anemia is a bone marrow failure syndrome characterized by and empty bone marrow and low blood counts. Most of the cases are immune-mediated. Allogeneic bone marrow transplant is the preferable treatment modality for patients younger than 40 years with a matched sibling donor. Patients not eligible for transplant are treated with intensive immunosuppressive therapy often based on anti-thymocyte globulin and cyclosporine.

However, up to one third of patients treated with immunosuppression are refractory and one third of those who response eventually relapse. Refractory and relapsed cases may be the result of insufficient immunosuppression and these cases may benefit from additional immunosuppression. Mesenchymal stem cells infusion may be a potential treatment option, considering its properties to modulate the immune system.

Refractory or relapsed patients with aplastic anemia will be treated with conventional immunosuppressive regimen (anti-thymocyte globulin plus cyclosporine) combined with intravenous infusion of allogeneic unrelated bone marrow mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acquired Aplastic Anemia
* Relapse/refractory to at least 1 immunosuppressive first line treatment
* Not eligible to allogeneic bone marrow transplantation

Exclusion Criteria:

* Previous or current malignancy
* Active or latent infectious disease
* Positive serologic tests for HIV, HCV, HBV, HTLV-1 and 2, Syphilis or Chagas disease
* Previous drug reaction for antithymocyte globulin, cyclosporin or corticosteroids
* Severe organic impairment (renal, hepatic, cardiac, pulmonary)
* Uncontrolled hypertension or diabetes
* Pregnancy
* Previous history of allergic reaction to penicillin or streptomycin
* Severe psychiatric disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of intravenous allogeneic unrelated mesenchymal stem cells infusion in patients with severe acquired aplastic anemia. | After the mesenchymal stem cells infusion up to 6 mounth after
  Adverse events like allergic reactions,infectious diseases,organ dysfunction or other related to mesenchymal stem cells infusion will be assessed.

SECONDARY OUTCOMES:
Level of cytopenias | weekly until 6 months
Transfusional requirements | weekly until 6 months
  Units of blood or platelets transfused after the mesenchymal stem cells infusion will be measured and compared to previously.
Incidence of infections and febrile neutropenia | weekly until 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Diego V Clé, MD, Principal Investigator — University of Sao Paulo; Rodrigo T Calado, MD, Study Chair — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Fouillard L, Bensidhoum M, Bories D, Bonte H, Lopez M, Moseley AM, Smith A, Lesage S, Beaujean F, Thierry D, Gourmelon P, Najman A, Gorin NC. Engraftment of allogeneic mesenchymal stem cells in the bone marrow of a patient with severe idiopathic aplastic anemia improves stroma. Leukemia. 2003 Feb;17(2):474-6. doi: 10.1038/sj.leu.2402786. No abstract available. PMID 12592355
- [Derived] Cle DV, Santana-Lemos B, Tellechea MF, Prata KL, Orellana MD, Covas DT, Calado RT. Intravenous infusion of allogeneic mesenchymal stromal cells in refractory or relapsed aplastic anemia. Cytotherapy. 2015 Dec;17(12):1696-705. doi: 10.1016/j.jcyt.2015.09.006. PMID 26589752